CLINICAL TRIAL: NCT03451851
Title: A Phase 3, Multicenter, Randomized, Placebo- and Active Comparator-Controlled Study Evaluating the Efficacy, Safety, and Pharmacokinetics of Subcutaneously Administered Guselkumab for the Treatment of Chronic Plaque Psoriasis in Pediatric Subjects (>=6 To <18 Years of Age)
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Subcutaneously Administered Guselkumab for the Treatment of Chronic Plaque Psoriasis in Pediatric Participants
Acronym: PROTOSTAR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR108452; CNTO1959PSO3011 (Other: Janssen Research & Development, LLC); 2023-503378-19-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — guselkumab; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 Group 1: Guselkumab (Experimental): Participants in Part 1a (age greater than or equal to (>=) 12 - less than (<) 18 years) will receive a weight-based dose of guselkumab subcutaneously (SC) at Weeks 0, 4, and 12. Participants who are PASI 90 responders at Week 16 will not receive any additional doses of guselkumab until they lose >=50% of their Week 16 PASI response, then they receive 1 dose guselkumab, followed by a dose 4 weeks later, and every 8 weeks (q8w) thereafter through Week 52. Participants who are PASI 90 non-responders at Week 16 will receive a placebo injection at Week 16 and continue to receive guselkumab q8w from Week 20 through Week 52. Participants who are eligible and willing to continue guselkumab may enter the Long Term Extension (LTE) Phase of the study. Part 1b (age >= 6 - <12 years) will follow the same dosing and commence after Part 1a data review.
  Interventions: Drug: Guselkumab; Drug: Placebo for guselkumab
- Part 1 Group 2: Placebo for Guselkumab (Placebo Comparator): Participants in Part 1a (age >= 12 - <18 years) will receive placebo for guselkumab administered SC at Weeks 0, 4, and 12. Participants who are PASI 90 responders at Week 16 will not receive any additional doses of study intervention until they lose >=50% of their Week 16 PASI response, at which time they will receive a weight-based guselkumab SC dose, followed by a dose 4 weeks later, and q8w thereafter through Week 52. Participants who are PASI 90 non-responders at Week 16 will receive a weight-based guselkumab dose at Weeks 16 and 20, followed by q8w dosing thereafter through Week 52. Participants who are eligible and willing to continue guselkumab treatment, may enter the LTE phase of the study. Part 1b (age >= 6 - <12 years) will follow the same dosing and commence after Part 1a data review.
  Interventions: Drug: Guselkumab; Drug: Placebo for guselkumab
- Part 1 Group 3: Etanercept (Active Comparator): Participants in Part 1a (age >= 12 - <18 years) will receive weight-based etanercept dose up to 50 milligram SC weekly through Week 15. Participants who elect to continue in the study will receive a weight-based guselkumab dose at Weeks 20 and 24, followed by q8w dosing thereafter through Week 48. Participants who are eligible and willing to continue guselkumab treatment, may enter the LTE phase of the study. Part 1b (age >= 6 - <12 years) will follow the same dosing and commence after Part 1a data review.
  Interventions: Drug: Guselkumab; Drug: Etanercept
- Part 2: Guselkumab (Experimental): Participants will receive a weight-based dose of open-label guselkumab SC at Weeks 0, 4 and q8w thereafter through Week 52. Participants who are eligible and willing to continue guselkumab treatment, may enter the LTE of the study and continue to receive guselkumab at Week 52 and q8w thereafter.
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Participants will receive a weight-based dose of guselkumab subcutaneously.
  Other Names: CNTO1959
Drug: Placebo for guselkumab — Participants will receive a weight-based dose of placebo for guselkumab subcutaneously.
  Arms: Part 1 Group 1: Guselkumab; Part 1 Group 2: Placebo for Guselkumab
Drug: Etanercept — Participants will receive a weight-based dose of etanercept (up to 50 mg) subcutaneously.
  Other Names: Enbrel
  Arms: Part 1 Group 3: Etanercept

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of guselkumab in pediatric participants aged greater than or equal to 6 through less than 18 years with chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of chronic plaque-type psoriasis for at least 6 months (with or without psoriatic arthritis [PsA]), prior to first administration of study intervention, defined as having at screening and baseline, Investigator Global Assessment (IGA) greater than or equal to (>=) 3, Psoriasis Area and Severity Index (PASI) >=12, >=10% body surface area (BSA) involvement and at least one of the following: very thick lesions, clinically relevant facial, genital, or hand/ foot involvement, PASI>=20, >20% BSA involvement, or IGA=4
* Be a candidate for phototherapy or systemic treatment of plaque psoriasis (either naive or history of previous treatment)
* Have plaque psoriasis considered by the investigator as inadequately controlled with phototherapy and/or topical therapy after an adequate dose and duration of therapy
* Be considered, in the opinion of the investigator, a suitable candidate for etanercept therapy, according to their country's approved Enbrel product labeling
* Be otherwise healthy on the basis of physical examination, medical history, and vital signs performed at screening. Any abnormalities, must be consistent with the underlying illness in the study population and this determination must be recorded in the participant's source documents and initialed by the investigator
* Must have acceptable evidence of immunity to varicella and measles, mumps, and rubella (MMR), which includes any one of the following: documentation of age-appropriate vaccination that includes both doses of each vaccine (unless local guidelines specify otherwise) or documentation of past infection by a healthcare provider or in the absence of previous 2 criteria, participants must have positive protective antibody titers to these infection prior to the first administration of study intervention. For participants who have not completed the recommended vaccination schedule for varicella and MMR, and the subsequent vaccination falls within the next 4 years, an accelerated vaccination schedule must be completed prior to study enrollment if available and required or strongly recommended for the location. If varicella or MMR vaccines are utilized, it is necessary for 2 weeks to elapse between the vaccination and receipt of study intervention

Exclusion Criteria:

* Currently has nonplaque forms of psoriasis (example, erythrodermic, guttate, or pustular)
* Has current drug-induced psoriasis (example, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
* Has previously received guselkumab or etanercept
* Has a history of chronic or recurrent infectious disease, including but not limited to chronic renal infection, chronic chest infection (example, bronchiectasis), recurrent urinary tract infection (recurrent pyelonephritis or chronic non-remitting cystitis), fungal infection (mucocutaneous candidiasis), or open, draining, or infected skin wounds or ulcers
* Has a known history of lymphoproliferative disease, including lymphoma; a history of monoclonal gammopathy of undetermined significance (MGUS); or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy or splenomegaly

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2026-12-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (39):
- United States (10):
  - Stanford University, Palo Alto, California
  - University of California, San Diego, San Diego, California
  - Dermatologic Surgery Specialists, Macon, Georgia
  - Northwestern University Feinberg School of Medicine Ann & Robert H Lurie Children's Hospital, Chicago, Illinois
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Windsor Dermatology, East Windsor, New Jersey
  - Mt. Sinai School of Medicine, New York, New York
  - Wright State Physicians Health Center, Dayton, Ohio
  - Arlington Center for Dermatology, Arlington, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
- Australia (3):
  - Eastern Health Research, Box Hill
  - Royal North Shore Hospital, St Leonards
  - Veracity Clinical Research, Woolloongabba
- Belgium (3):
  - Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Centre Hospitalier Universitaire de Liege Domaine Universitaire du Sart Tilman, Liège
- Canada (3):
  - Kirk Barber Reseach Inc., Calgary, Alberta
  - Dermatology Research Institute Inc, Calgary, Alberta
  - Skin Care Centre, Vancouver, British Columbia
- Germany (7):
  - Universitatsklinikum Bonn, Bonn
  - Universitatsklinikum Carl Gustav Carcus Dresden, Dresden
  - Universitatsklinikum Frankfurt, Frankfurt
  - Universitatsklinikum Schleswig Holstein Kiel, Kiel
  - Praxis Dr. med. Beate Schwarz - Germany, Langenau
  - Company for Medical Study & Service Selters, Selters
  - Hautarztpraxis Dr. Leitz & Kollegen, Stuttgart
- Hungary (4):
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Debreceni Egyetem, Debrecen
  - Borsod Abauj Zemplen Varmegyei Kozponti Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Szegedi Tudomanyegyetem, Szeged
- Italy (5):
  - Ospedali Riuniti Di Ancona, Ancona
  - Azienda Ospedaliera Policlinico S. Orsola-Malpighi, Bologna
  - AOU di Cagliari, Cagliari
  - Azienda Ospedaliera di Padova, Padua
  - Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia
- Radboud University Medical Center, Nijmegen, Netherlands
- Poland (3):
  - Dermed Centrum Medyczne Sp z o o, Lodz
  - Szpital Dzieciecy im. prof. dr. med. Jana Bogdanowicza w Warszawie, Warsaw
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw

REFERENCES:
- [Derived] Crauwels H, Ringold S, Howard S, Van Hartingsveldt B, Smith V, Jett M, Baguet T, Adamson E, Chakravarty SD, Leu JH. Extrapolating Guselkumab Efficacy to Juvenile Psoriatic Arthritis from Adult Psoriatic Arthritis and Adult and Pediatric Psoriasis Data. Paediatr Drugs. 2025 Oct 28. doi: 10.1007/s40272-025-00725-2. Online ahead of print. PMID 41152645
- [Derived] Prajapati VH, Seyger MMB, Wilsmann-Theis D, Szakos E, Kaszuba A, van Hartingsveldt B, Jett M, Jiang G, Li S, Sinha V, Crauwels H, DeKlotz CMC, Paller AS. Guselkumab for the treatment of moderate-to-severe plaque psoriasis in paediatric patients: results of the phase III randomized placebo-controlled PROTOSTAR study. Br J Dermatol. 2025 Mar 18;192(4):618-628. doi: 10.1093/bjd/ljae502. PMID 39708367

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This result is currently reported for primary analysis till clinical cut-off date 29-Mar-2024. In Part 1, the enrollment of participants aged greater than or equal to (>=) 6 to less than (<) 12 years started only after all participants aged >=12 to <18 years of age had finished Week 16 of the study. Long-term extension (LTE) phase is still ongoing, and results will be posted upon study completion.
Groups:
- Group 1 (Part 1): Placebo (Week 0-16): Adolescent participants (aged >=12 to <18 years) received placebo matched to guselkumab as subcutaneous (SC) injection at Weeks 0, 4, and 12 during the placebo-controlled period (PCP). Once adolescent participants completed Week 16, eligible participants aged >=6 to <12 years were enrolled and began receiving the same dose regimen starting from Week 0 until Week 16.
- Group 2 (Part 1): Guselkumab (Week 0-16): Adolescent participants received weight-adjusted doses of guselkumab (1.3 mg/kg for body weight [BW] <70 kg, 100 mg for BW >=70 kg) via subcutaneous injection at Weeks 0, 4, and 12 during PCP. Once adolescent participants completed Week 16, eligible participants aged >=6 to <12 years began receiving the same dose regimen starting from Week 0 until Week 16.
- Group 3 (Part 1): Etanercept (Week 0-16): Adolescent participants received weight-based dose of open-label etanercept 0.8 mg/kg for BW <63 kg and 50 mg for BW >=63 kg SC injection once weekly from Week 0 to Week 15. Once adolescent participants completed Week 16, eligible participants aged >=6 to <12 years began receiving the same dose regimen starting from Week 0 until Week 16.
- Group 1 (Part 1): Placebo to Guselkumab (Week 16-52): Participants who received placebo during PCP were assessed for psoriasis area and severity index (PASI) response at Week 16. Participants who were PASI 90 non-responders at Week 16 received weight-based doses of guselkumab (1.3 mg/kg for BW <70 kg, 100 mg for BW >=70 kg) as SC injection at Weeks 16, 20 and then every 8 weeks (q8w) thereafter through Week 52. Participants who were PASI 90 responders at Week 16 stopped treatment until they lost >= 50 percent (%) of their Week 16 PASI response, at which time they were treated with guselkumab 1.3 mg/kg or 100 mg depending on their body weight followed by a dose 4 weeks later, and then guselkumab q8w thereafter through Week 52. All participants who completed Part 1 of the main study through Week 52 were offered the opportunity to participate in an open-label LTE.
- Group 2 (Part 1): Guselkumab (Week 16-52): Participants who received guselkumab during PCP were assessed for PASI response at Week 16. Participants who were PASI 90 non-responders at Week 16 received weight-based doses of guselkumab (1.3 mg/kg for BW <70 kg, 100 mg for BW >=70 kg) as SC injection at Weeks 16, 20 and then q8w thereafter through Week 52. Participants who were PASI 90 responders at Week 16 stopped treatment until they lost >= 50 % of their Week 16 PASI response, at which time they were retreated with guselkumab 1.3 mg/kg or 100 mg depending on their body weight followed by a dose 4 weeks later, and then guselkumab every 8 weeks thereafter through Week 52. All participants who completed Part 1 of the main study through Week 52 were offered the opportunity to participate in an open-label LTE.
- Group 3 (Part 1): Etanercept to Guselkumab (Week 16-52): Participants who received etanercept during the PCP had the option to continue in the study or to discontinue the study. Participants that continued received weight-based doses of guselkumab (1.3 mg/kg for body weight [BW] <70 kg, 100 mg for BW >=70 kg) as SC injection at Weeks 20 and 24, followed by q8w dosing through Week 48 and remaining participants discontinued from the study. All participants who completed Part 1 of the main study through Week 52 were offered the opportunity to participate in an open-label LTE.
- Part 2: Guselkumab (Week 0-16): Adolescent participants received weight-based dose of open-label guselkumab (1.3 mg/kg for body weight [BW] <70 kg, 100 mg for BW >=70 kg) as SC injection at Weeks 0, 4, and 16.
- Part 2: Guselkumab (Week 16-52): Participants who completed Week 16 during PCP continued to receive weight-based dose of open-label guselkumab (1.3 mg/kg for body weight [BW] <70 kg, 100 mg for BW >=70 kg) as SC injection q8w from Weeks 16 through Week 52. All participants who completed Part 2 of the main study through Week 52 were offered the opportunity to participate in an open-label LTE.
Period: PCP: Week 0 -16
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16) | Group 1 (Part 1): Placebo to Guselkumab (Week 16-52) | Group 2 (Part 1): Guselkumab (Week 16-52) | Group 3 (Part 1): Etanercept to Guselkumab (Week 16-52) | Part 2: Guselkumab (Week 0-16) | Part 2: Guselkumab (Week 16-52)
Started | 25 | 41 | 26 | 0 | 0 | 0 | 28 | 0
Completed | 24 | 41 | 23 | 0 | 0 | 0 | 27 | 0
Not Completed | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Period: Withdrawal and Retreament: Week 16-52
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16) | Group 1 (Part 1): Placebo to Guselkumab (Week 16-52) | Group 2 (Part 1): Guselkumab (Week 16-52) | Group 3 (Part 1): Etanercept to Guselkumab (Week 16-52) | Part 2: Guselkumab (Week 0-16) | Part 2: Guselkumab (Week 16-52)
Started | 0 | 0 | 0 | 23 (Only eligible participants who crossed over to receive Guselkumab included in this period.) | 41 | 22 (Only eligible participants who crossed over to receive Guselkumab included in this period.) | 0 | 27
Completed | 0 | 0 | 0 | 23 | 35 | 21 | 0 | 27
Not Completed | 0 | 0 | 0 | 0 | 6 | 1 | 0 | 0
Not completed — Other Withdrawal by Parent/Guardian | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Not completed — Other Unspecified | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other- completed safety follow up | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16) | Part 2: Guselkumab (Week 0-16) | Total
Number analyzed (Participants) | 25 | 41 | 26 | 28 | 120
Age, Customized [Count of Participants; unit: Participants]
  >=6 to <12 years | 10 | 10 | 10 | 0 | 30
  >=12 to <18 years | 15 | 31 | 16 | 28 | 90
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 11 | 11 | 52
  Male | 12 | 24 | 15 | 17 | 68
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 2 | 0 | 4
  Black or African American | 2 | 1 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 20 | 36 | 22 | 28 | 106
  More than one race | 0 | 1 | 1 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
  Other | 1 | 2 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  AUSTRALIA | 0 | 1 | 0 | 0 | 1
  BELGIUM | 0 | 4 | 5 | 2 | 11
  CANADA | 1 | 5 | 1 | 1 | 8
  GERMANY | 4 | 4 | 5 | 9 | 22
  HUNGARY | 6 | 11 | 4 | 9 | 30
  ITALY | 4 | 4 | 1 | 1 | 10
  NETHERLANDS | 1 | 2 | 0 | 0 | 3
  POLAND | 5 | 7 | 6 | 6 | 24
  UNITED STATES | 4 | 3 | 4 | 0 | 11
AgeContinuous [Mean (Standard Deviation); unit: years] | 12.4 (3.63) | 13.4 (2.86) | 12.5 (3.29) | 15.1 (1.59) | 13.4 (3.05)

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants Who Achieved an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) at Week 16
Description: The IGA assesses participant's plaque psoriasis. Lesions were graded for induration, erythema and scaling, each using a 5 point scale. Induration: 0 = no evidence of plaque elevation, 1 = minimal plaque elevation, = 0.25 mm; 2 = mild plaque elevation, = 0.5 mm; 3 = moderate plaque elevation, = 0.75 mm; 4 = severe plaque elevation, >1 mm; Erythema: 0 = no evidence of erythema, hyperpigmentation may be present, 1 = faint erythema, 2 = light red coloration, 3 = moderate red coloration, 4 = bright red coloration; Scaling: 0 = no evidence of scaling, 1 = minimal; occasional fine scale over less than 5% of the lesion, 2 = mild; fine scale dominates, 3 = moderate; coarse scale predominates, 4 = severe; thick, scale predominates. Final IGA score of psoriasis was based upon the average of induration, erythema and scaling scores assessed on a 5 point scale: cleared (0), minimal (1), mild (2), moderate (3), or severe (4). A higher score indicated more severe disease.
Time Frame: At Week 16
Population: The efficacy analysis for Part 1 of the study was based upon the full analysis set (FAS) which included all randomized participants in Part 1. In the efficacy analyses, participants were analyzed according to their assigned treatment group regardless of their actual treatment received.
Measure: Number; unit: Percentages of participants
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16)
Number analyzed (Participants) | 25 | 41 | 26
Percentages of participants | 16.0 | 65.9 | 69.2
Statistical Analysis 1: Comparison: Group 1 (Part 1): Placebo (Week 0-16) vs Group 2 (Part 1): Guselkumab (Week 0-16); Guselkumab Vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact; P-values represented the comparisons with placebo and were based on the Fisher's exact test stratified by age group and region (pooled); Difference in percentage = 49.9, 95% CI 2-sided [25.9 to 69.4]

2. Primary Outcome: Part 1: Percentage of Participants Who Achieved Psoriasis Area and Severity Index (PASI) 75 Response at Week 16
Description: The PASI was a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body was divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produced a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicated more severe disease. A PASI 75 response represented participants who achieved at least a 75 % improvement from baseline in the PASI score.
Time Frame: At Week 16
Population: The efficacy analysis for Part 1 of the study was based upon the FAS which included all randomized participants in Part 1. In the efficacy analyses, participants were analyzed according to their assigned treatment group regardless of their actual treatment received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16)
Number analyzed (Participants) | 25 | 41 | 26
Percentage of Participants | 20.0 | 75.6 | 69.2
Statistical Analysis 1: Comparison: Group 1 (Part 1): Placebo (Week 0-16) vs Group 2 (Part 1): Guselkumab (Week 0-16); Guselkumab Vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact; [statistical method as in outcome 1, analysis 1]; Difference in percentage = 55.6, 95% CI 2-sided [32.1 to 74.0]

3. Secondary Outcome: Part 1: Percentage of Participants Who Achieve PASI 90 Response at Week 16
Description: The PASI was a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body was divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 % to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produced a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicated more severe disease. A PASI 90 response represented participants who achieved at least a 90 % improvement from baseline in the PASI score.
Time Frame: At Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16)
Number analyzed (Participants) | 25 | 41 | 26
Percentage of Participants | 16.0 | 56.1 | 53.8
Statistical Analysis 1: Comparison: Group 1 (Part 1): Placebo (Week 0-16) vs Group 2 (Part 1): Guselkumab (Week 0-16); Guselkumab Vs Placebo; Test type: Superiority; p = 0.003, Fisher Exact; [statistical method as in outcome 1, analysis 1]; Difference in percentage = 40.1, 95% CI 2-sided [15.6 to 61.3]

4. Secondary Outcome: Part 1: Percentage of Participants Who Achieved an IGA Score of Cleared (0) at Week 16
Description: as for outcome 1
Time Frame: At Week 16
Population: as for outcome 2
Measure: Number; unit: Percentages of participants
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16)
Number analyzed (Participants) | 25 | 41 | 26
Percentages of participants | 4.0 | 39.0 | 26.9
Statistical Analysis 1: Comparison: Group 1 (Part 1): Placebo (Week 0-16) vs Group 2 (Part 1): Guselkumab (Week 0-16); Guselkumab Vs Placebo; Test type: Superiority; p = 0.004, Fisher Exact; [statistical method as in outcome 1, analysis 1]; Difference in percentage = 35, 95% CI 2-sided [10.5 to 56.8]

5. Secondary Outcome: Part 1: Percentage of Participants Who Achieved PASI 100 Response at Week 16
Description: The PASI was a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body was divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent [%] to 100% involvement), and for erythema, induration, and scaling, which were each rated on a scale of 0 (none) to 4 (severe). The PASI produced a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicated more severe disease. A PASI 100 response represented participants who achieved a 100 % improvement from baseline in the PASI score.
Time Frame: At Week 16
Population: as for outcome 2
Measure: Number; unit: Percentages of participants
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16)
Number analyzed (Participants) | 25 | 41 | 26
Percentages of participants | 0 | 34.1 | 26.9
Statistical Analysis 1: Comparison: Group 1 (Part 1): Placebo (Week 0-16) vs Group 2 (Part 1): Guselkumab (Week 0-16); Guselkumab Vs Placebo; Test type: Superiority; p = 0.002, Fisher Exact; [statistical method as in outcome 1, analysis 1]; Difference in percentage = 34.1, 25% CI 2-sided [9.7 to 56.1]

6. Secondary Outcome: Part 1: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) Score at Week 16
Description: CDLQI is a 10-item questionnaire that measures the impact of skin disease on children's quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. CDLQI total score was the sum of individual scores of questions 1-10 and ranged from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of children. Change from baseline is defined as post baseline score minus baseline score.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16)
Number analyzed (Participants) | 25 | 41 | 26
Score on a scale | -1.68 (6.323) | -7.12 (7.633) | -6.08 (5.692)
Statistical Analysis 1: Comparison: Group 1 (Part 1): Placebo (Week 0-16) vs Group 2 (Part 1): Guselkumab (Week 0-16); Guselkumab Vs Placebo; Test type: Superiority; p < 0.001, Mixed model repeated measures (MMRM); LS Mean difference = -5.4, 95% CI 2-sided [-7.33 to -3.06]

7. Secondary Outcome: Part 1: Percentage of Retreated Participants Who Achieved a PASI 90 Response Over Time After Retreatment
Description: PASI was a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In PASI system, body was divided into 4 regions: head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for percentage of area involved, which translates to score that ranges from 0 (indicates no involvement) to 6 (90 % to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). PASI produced a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicated more severe disease. A PASI 90 response represented participants who achieved at least a 90 % improvement from baseline in PASI score.
Time Frame: At 4 and 8 weeks post retreatment (retreatment period ranged from Week 16 to Week 52)
Population: Analysis population included Guselkumab PASI 90 responders at Week 16 who were retreated with guselkumab prior to Week 52. This outcome measure was planned to be analyzed for "Group 2 (Part 1): Guselkumab (Week 16-52)" arm only. Here, n (Number Analyzed) signifies number of participants evaluable at specified time points.
Measure: Number; unit: Percentages of participants
Arm/Group | Group 2 (Part 1): Guselkumab (Week 16-52)
Number analyzed (Participants) | 4
Percentages of participants
  4 weeks after retreatment of guselkumab | 0
  8 weeks after retreatment of guselkumab: number analyzed (Participants) | 2
  8 weeks after retreatment of guselkumab | 50.0

8. Secondary Outcome: Part 1: Percentage of Retreated Participants Who Achieved PASI Responses (PASI 50, 75, 90, and 100) Over Time After Retreatment
Description: The PASI was a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body was divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produced a numeric score that can range from 0 (no psoriasis) to 72. A higher score indicated more severe disease. PASI 50, 75, 90 and 100 response represented at least 50, 75, 90 and 100% improvement from baseline respectively, in the PASI score.
Time Frame: At 4 and 8 weeks post retreatment (retreatment period ranged from Week 16 to Week 52)
Population: Analysis population included guselkumab PASI 90 responders at Week 16 who were retreated with guselkumab prior to Week 52. Here, n (Number Analyzed) signifies number of participants evaluable at specified time points. This outcome measure was planned to be analyzed for "Group 2 (Part 1): Guselkumab (Week 16-52)" arm only.
Measure: Number; unit: At 4 and 8 weeks post retreatment
Arm/Group | Group 2 (Part 1): Guselkumab (Week 16-52)
Number analyzed (Participants) | 4
At 4 and 8 weeks post retreatment
  4 weeks after retreatment: >=50% improvement | 50.0
  4 weeks after retreatment: >=75% improvement | 0
  4 weeks after retreatment:>= 90% improvement | 0
  4 weeks after retreatment: 100% improvement | 0
  8 weeks after retreatment: >=50% improvement: number analyzed (Participants) | 2
  8 weeks after retreatment: >=50% improvement | 50.0
  8 weeks after retreatment: >=75% improvement: number analyzed (Participants) | 2
  8 weeks after retreatment: >=75% improvement | 50.0
  8 weeks after retreatment:>= 90% improvement: number analyzed (Participants) | 2
  8 weeks after retreatment:>= 90% improvement | 50.0
  8 weeks after retreatment: 100% improvement: number analyzed (Participants) | 2
  8 weeks after retreatment: 100% improvement | 50.0

9. Secondary Outcome: Part 1: Percentage of Retreated Participants Who Achieved IGA Responses (IGA of Cleared [0], Minimal [1], or Mild [2], IGA of Cleared [0] or Minimal [1], and IGA of Cleared [0]) Over Time After Retreatment
Description: The IGA assesses participant's plaque psoriasis. Lesions were graded for induration, erythema and scaling, each using a 5 points scale. Induration: 0 = no evidence of plaque elevation, 1 = minimal plaque elevation, = 0.25 mm; 2 = mild plaque elevation, = 0.5 mm; 3 = moderate plaque elevation, = 0.75 mm; 4 = severe plaque elevation, >1 mm; Erythema: 0 = no evidence of erythema, hyperpigmentation may be present, 1 = faint erythema, 2 = light red coloration, 3 = moderate red coloration, 4 = bright red coloration; Scaling: 0 = no evidence of scaling, 1 = minimal; occasional fine scale over less than 5% of the lesion, 2 = mild; fine scale dominates, 3 = moderate; coarse scale predominates, 4 = severe; thick, scale predominates. Final IGA score of psoriasis was based upon the average of induration, erythema and scaling scores assessed on a 5 points scale: cleared (0), minimal (1), mild (2), moderate (3), or severe (4). A higher score indicated more severe disease.
Time Frame: At 4 and 8 weeks post retreatment (retreatment period ranged from Week 16 to Week 52)
Population: as for outcome 8
Measure: Number; unit: Percentages of participants
Arm/Group | Group 2 (Part 1): Guselkumab (Week 16-52)
Number analyzed (Participants) | 4
Percentages of participants
  4 Weeks after retreatment: IGA-0 | 0
  4 Weeks after retreatment: IGA-0 or 1 | 25.0
  4 Weeks after retreatment: IGA-2 | 75.0
  8 Weeks after retreatment: IGA-0: number analyzed (Participants) | 2
  8 Weeks after retreatment: IGA-0 | 50.0
  8 Weeks after retreatment: IGA-0 or 1: number analyzed (Participants) | 2
  8 Weeks after retreatment: IGA-0 or 1 | 50.0
  8 Weeks after retreatment: IGA- 2: number analyzed (Participants) | 2
  8 Weeks after retreatment: IGA- 2 | 100.0

10. Secondary Outcome: Part 1: Cumulative Rate of Loss of at Least 50% of Week 16 PASI Improvement Through Week 52 Among Guselkumab PASI 90 Responders at Week 16
Description: Cumulative rate of loss of at least 50% of PASI improvement was defined as percentage of participants with a loss of >=50% of Week 16 PASI improvement after treatment is withdrawn. The PASI was a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In PASI system, body was divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 % to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produced a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicated more severe disease.
Time Frame: Weeks 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Analysis population included Guselkumab PASI 90 responders at Week 16. This outcome measure was planned to be analyzed for "Group 2 (Part 1): Guselkumab (Week 16-52)" arm only.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 2 (Part 1): Guselkumab (Week 16-52)
Number analyzed (Participants) | 23
Percentage of Participants
  Week 20 | 0
  Week 24 | 0
  Week 28 | 0
  Week 32 | 0
  Week 36 | 0
  Week 40 | 0
  Week 44 | 9.3
  Week 48 | 19.1
  Week 52 | 19.1

11. Secondary Outcome: Part 1: Cumulative Maintenance Rate of PASI 90 Response Through Week 52 Among Guselkumab PASI 90 Responders at Week 16
Description: Cumulative maintenance rate was defined as percentage of participants who maintained their PASI 90 response through Week 52 among guselkumab PASI 90 responders at Week 16. The PASI was a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In PASI system, body was divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produced a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicated more severe disease. A PASI 90 response represented participants who achieved at least a 90% improvement from baseline in PASI score.
Time Frame: Week 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Group 2 (Part 1): Guselkumab (Week 16-52)
Number analyzed (Participants) | 23
Percentage of participants
  Week 20 | 100
  Week 24 | 100
  Week 28 | 86.7
  Week 32 | 77.5
  Week 36 | 63.9
  Week 40 | 50.2
  Week 44 | 35.8
  Week 48 | 30.7
  Week 52 | 25.6

12. Secondary Outcome: Part 1: Percentage of Participants Who Achieved a PASI 50 Response at Week 16
Description: The PASI was a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. The PASI was a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In PASI system, body was divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 % to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produced a numeric score that can range from 0 (no visible skin involvement) to 72 (maximal skin involvement of the whole body). A higher score indicated more severe disease. A PASI 50 response represented at least a 50% improvement from baseline in the PASI score.
Time Frame: At Week 16
Population: as for outcome 2
Measure: Number; unit: Percentages of participants
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16)
Number analyzed (Participants) | 25 | 41 | 26
Percentages of participants | 28.0 | 87.8 | 76.9
Statistical Analysis 1: Comparison: Group 1 (Part 1): Placebo (Week 0-16) vs Group 2 (Part 1): Guselkumab (Week 0-16); Guselkumab Vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — p-value is nominal; [statistical method as in outcome 1, analysis 1]; Difference in percentage = 59.8, 95% CI 2-sided [36.9 to 77.6]

13. Secondary Outcome: Part 1: Percent Improvement From Baseline in PASI Through Week 16
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body was divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produced a numeric score that can range from 0 (no psoriasis) to 72. A higher score indicated more severe disease.
Time Frame: Weeks 4, 8, 12, and 16
Population: The efficacy analysis for Part 1 of the study was based upon the FAS which included all randomized participants in Part 1. In the efficacy analyses, participants were analyzed according to their assigned treatment group regardless of their actual treatment received. Here, n (number analyzed): number of participants evaluable for each arm at specified time points.
Measure: Mean (Standard Deviation); unit: Percent improvement
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16)
Number analyzed (Participants) | 25 | 41 | 26
Percent improvement
  Week 4: number analyzed (Participants) | 25 | 41 | 25
  Week 4 | 13.37 (30.074) | 39.12 (27.907) | 42.53 (26.013)
  Week 8: number analyzed (Participants) | 24 | 39 | 26
  Week 8 | 13.61 (40.734) | 71.25 (28.018) | 64.27 (29.314)
  Week 12: number analyzed (Participants) | 25 | 41 | 24
  Week 12 | 13.67 (52.391) | 79.79 (28.570) | 77.30 (24.735)
  Week 16: number analyzed (Participants) | 25 | 41 | 24
  Week 16 | 16.02 (55.538) | 79.83 (30.468) | 82.05 (23.225)

14. Secondary Outcome: Part 2: Percent Improvement From Baseline in PASI Through Week 52
Description: The PASI was a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body was divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which were each rated on a scale of 0 to 4. The PASI produced a numeric score that can range from 0 (no psoriasis) to 72. A higher score indicated more severe disease.
Time Frame: Weeks 4, 8, 12, 16, 20, 28, 36, 44, and 52
Population: FAS for Part 2 included all participants enrolled in Part 2. Here, n (number analyzed) signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Percent improvement
Groups:
- Part 2: Guselkumab (Week 0-52): Adolescent participants received weight-based dose of open-label guselkumab (1.3 mg/kg for body weight [BW] <70 kg, 100 mg for BW >=70 kg) as SC injection at Weeks 0, 4, and q8w thereafter through Week 52. All participants who completed Part 2 of the main study through Week 52 were offered the opportunity to participate in an open-label LTE.
Arm/Group | Part 2: Guselkumab (Week 0-52)
Number analyzed (Participants) | 28
Percent improvement
  Week 4 | 48.33 (26.781)
  Week 8 | 79.05 (21.177)
  Week 12: number analyzed (Participants) | 27
  Week 12 | 86.40 (15.541)
  Week 16: number analyzed (Participants) | 26
  Week 16 | 91.96 (11.177)
  Week 20: number analyzed (Participants) | 27
  Week 20 | 91.10 (14.851)
  Week 28: number analyzed (Participants) | 27
  Week 28 | 93.44 (12.948)
  Week 36: number analyzed (Participants) | 27
  Week 36 | 95.77 (7.848)
  Week 44: number analyzed (Participants) | 27
  Week 44 | 95.95 (7.430)
  Week 52: number analyzed (Participants) | 27
  Week 52 | 96.32 (7.478)

15. Secondary Outcome: Part 1: Percentage of Participants With PASI Responses (PASI 50, 75, 90, and 100) Through Week 16
Description: The PASI was a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body was divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which were each rated on a scale of 0 to 4. The PASI produced a numeric score that can range from 0 (no psoriasis) to 72. A higher score indicated more severe disease. PASI 50, 75, 90, and 100 responses represented at least 50%, 75%, 90%, and 100% improvement from baseline respectively, in the PASI score.
Time Frame: Weeks 4, 8, 12, and 16
Population: as for outcome 2
Measure: Number; unit: Percentages of participants
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16)
Number analyzed (Participants) | 25 | 41 | 26
Percentages of participants
  Week 4: >= 50% improvement | 8.0 | 34.1 | 38.5
  Week 4: >= 75% improvement | 8.0 | 12.2 | 15.4
  Week 4: >= 90% improvement | 4.0 | 2.4 | 3.8
  Week 4: 100% improvement | 0 | 0 | 0
  Week 8: >= 50% improvement | 20.0 | 78.0 | 73.1
  Week 8: >= 75% improvement | 8.0 | 51.2 | 46.2
  Week 8: >= 90% improvement | 4.0 | 34.1 | 19.2
  Week 8: 100% improvement | 4.0 | 12.2 | 11.5
  Week 12: >= 50% improvement | 24.0 | 85.4 | 76.9
  Week 12: >= 75% improvement | 12.0 | 73.2 | 61.5
  Week 12: >= 90% improvement | 8.0 | 56.1 | 38.5
  Week 12: 100% improvement | 0 | 34.1 | 26.9
  Week 16: >= 50% improvement | 28.0 | 87.8 | 76.9
  Week 16: >= 75% improvement | 20.0 | 75.6 | 69.2
  Week 16: >= 90% improvement | 16.0 | 56.1 | 53.8
  Week 16: 100% improvement | 0 | 34.1 | 26.9

16. Secondary Outcome: Part 2: Percentage of Participants With PASI Responses (PASI 50, 75, 90, and 100) Through Week 52
Description: The PASI was a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body was divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produced a numeric score that can range from 0 (no psoriasis) to 72. A higher score indicated more severe disease. PASI 50, 75, 90, and 100 responses represented at least 50%, 75%, 90%, and 100% improvement from baseline respectively, in the PASI score.
Time Frame: Weeks 4, 8, 12, 16, 20, 28, 36, 44, and 52
Population: FAS for Part 2 included all participants enrolled in Part 2.
Measure: Number; unit: Percentages of participants
Arm/Group | Part 2: Guselkumab (Week 0-52)
Number analyzed (Participants) | 28
Percentages of participants
  Week 4: >= 50% improvement | 42.9
  Week 4: >= 75% improvement | 14.3
  Week 4: >= 90% improvement | 14.3
  Week 4: 100% improvement | 3.6
  Week 8: >= 50% improvement | 89.3
  Week 8: >= 75% improvement | 67.9
  Week 8: >= 90% improvement | 39.3
  Week 8: 100% improvement | 17.9
  Week 12: >= 50% improvement | 96.4
  Week 12: >= 75% improvement | 75.0
  Week 12: >= 90% improvement | 42.9
  Week 12: 100% improvement | 25.0
  Week 16: >= 50% improvement | 92.9
  Week 16: >= 75% improvement | 82.1
  Week 16: >= 90% improvement | 64.3
  Week 16: 100% improvement | 35.7
  Week 20: >= 50% improvement | 92.9
  Week 20: >= 75% improvement | 82.1
  Week 20: >= 90% improvement | 75.0
  Week 20: 100% improvement | 39.3
  Week 28: >= 50% improvement | 92.9
  Week 28: >= 75% improvement | 89.3
  Week 28: >= 90% improvement | 75.0
  Week 28: 100% improvement | 46.4
  Week 36: >= 50% improvement | 96.4
  Week 36: >= 75% improvement | 89.3
  Week 36: >= 90% improvement | 82.1
  Week 36: 100% improvement | 53.6
  Week 44: >= 50% improvement | 96.4
  Week 44: >= 75% improvement | 89.3
  Week 44: >= 90% improvement | 82.1
  Week 44: 100% improvement | 53.6
  Week 52: >= 50% improvement | 96.4
  Week 52: >= 75% improvement | 92.9
  Week 52: >= 90% improvement | 82.1
  Week 52: 100% improvement | 53.6

17. Secondary Outcome: Part 1: Percentage of Participants With IGA of Cleared (0), Cleared (0) or Minimal (1), Mild or Better (<=2) Through Week 16
Description: as for outcome 9
Time Frame: Weeks 4, 8, 12, and 16
Population: as for outcome 2
Measure: Number; unit: Percentages of participants
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16)
Number analyzed (Participants) | 25 | 41 | 26
Percentages of participants
  Week 4 : IGA of cleared (0) | 0 | 0 | 0
  Week 4 : IGA of cleared (0) or minimal (1) | 8.0 | 19.5 | 23.1
  Week 4 :IGA of mild or better (<=2) | 20.0 | 63.4 | 73.1
  Week 8: IGA of cleared (0) | 4.0 | 22.0 | 11.5
  Week 8 : IGA of cleared (0) or minimal (1) | 8.0 | 58.5 | 50.0
  Week 8 :IGA of mild or better (<=2) | 24.0 | 78.0 | 88.5
  Week 12: IGA of cleared (0) | 4.0 | 43.9 | 26.9
  Week 12 : IGA of cleared (0) or minimal (1) | 8.0 | 70.7 | 65.4
  Week 12 :IGA of mild or better (<=2) | 40.0 | 87.8 | 84.6
  Week 16: IGA of cleared (0) | 4.0 | 39.0 | 26.9
  Week 16 : IGA of cleared (0) or minimal (1) | 16.0 | 65.9 | 69.2
  Week 16 :IGA of mild or better (<=2) | 48.0 | 92.7 | 84.6

18. Secondary Outcome: Part 2: Percentage of Participants With IGA of Cleared (0), Cleared (0) or Minimal (1), Mild or Better (<=2) Through Week 52
Description: as for outcome 9
Time Frame: Weeks 4, 8, 12, 16, 20, 28, 36, 44, and 52
Population: FAS for Part 2 included all participants enrolled in Part 2.
Measure: Number; unit: Percentages of participants
Arm/Group | Part 2: Guselkumab (Week 0-52)
Number analyzed (Participants) | 28
Percentages of participants
  Week 4: IGA of cleared (0) | 3.6
  Week 4: IGA of cleared (0) or minimal (1) | 25.0
  Week 4:IGA of mild or better (<=2) | 57.1
  Week 8: IGA of cleared (0) | 25.0
  Week 8: IGA of cleared (0) or minimal (1) | 64.3
  Week 8:IGA of mild or better (<=2) | 92.9
  Week 12: IGA of cleared (0) | 35.7
  Week 12: IGA of cleared (0) or minimal (1) | 75.0
  Week 12:IGA of mild or better (<=2) | 96.4
  Week 16: IGA of cleared (0) | 46.4
  Week 16: IGA of cleared (0) or minimal (1) | 89.3
  Week 16:IGA of mild or better (<=2) | 92.9
  Week 20: IGA of cleared (0) | 50.0
  Week 20: IGA of cleared (0) or minimal (1) | 82.1
  Week 20:IGA of mild or better (<=2) | 96.4
  Week 28: IGA of cleared (0) | 57.1
  Week 28: IGA of cleared (0) or minimal (1) | 78.6
  Week 28:IGA of mild or better (<=2) | 96.4
  Week 36: IGA of cleared (0) | 64.3
  Week 36: IGA of cleared (0) or minimal (1) | 89.3
  Week 36:IGA of mild or better (<=2) | 89.3
  Week 44: IGA of cleared (0) | 64.3
  Week 44: IGA of cleared (0) or minimal (1) | 85.7
  Week 44: IGA of mild or better (<=2) | 89.3
  Week 52: IGA of cleared (0) | 75.0
  Week 52: IGA of cleared (0) or minimal (1) | 85.7
  Week 52: IGA of mild or better (<=2) | 92.9

19. Secondary Outcome: Part 2: Change From Baseline in CDLQI Score Through Week 52
Description: Change from baseline in CDLQI score through Week 52 were reported. CDLQI is a 10-item questionnaire that measures the impact of skin disease on children's quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. CDLQI total score was the sum of individual scores of questions 1-10 and ranged from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of children.
Time Frame: Baseline, Weeks 8, 16, 28, 36, and 52
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part 2: Guselkumab (Week 0-52)
Number analyzed (Participants) | 28
Score on a scale
  Week 8 | -5.6 (6.40)
  Week 16: number analyzed (Participants) | 26
  Week 16 | -6.8 (6.32)
  Week 28: number analyzed (Participants) | 27
  Week 28 | -6.7 (6.54)
  Week 36: number analyzed (Participants) | 27
  Week 36 | -7.0 (6.88)
  Week 52: number analyzed (Participants) | 26
  Week 52 | -7.3 (6.83)

20. Secondary Outcome: Part 1: Percentage of Participants With CDLQI Score Equal to 0 or 1 at Week 16 Among Participants With a Baseline CDLQI Score Greater Than (>) 1
Description: CDLQI is a 10-item questionnaire that measures the impact of skin disease on children's quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. CDLQI total score was the sum of individual scores of question 1-10 and ranges from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of children.
Time Frame: At Week 16
Population: The efficacy analysis for Part 1 of the study was based upon the FAS which included all randomized participants in Part 1. In the efficacy analyses, participants were analyzed according to their assigned treatment group regardless of their actual treatment received. Here, N (Overall Number of Participants Analyzed) signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentages of participants
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16)
Number analyzed (Participants) | 23 | 39 | 26
Percentages of participants | 17.4 | 64.1 | 38.5
Statistical Analysis 1: Comparison: Group 1 (Part 1): Placebo (Week 0-16) vs Group 2 (Part 1): Guselkumab (Week 0-16); Test type: Superiority; p = 0.002, Fisher Exact — p-value is nominal; [statistical method as in outcome 1, analysis 1]; Difference in percentage = 46.7, 95% CI 2-sided [21.9 to 67.3]

21. Secondary Outcome: Part 2: Percentage of Participants With CDLQI Score Equal to of 0 or 1 Through Week 52 Among Participants With a Baseline CDLQI Score > 1
Description: as for outcome 20
Time Frame: Weeks 8, 16, 28, 36, and 52
Population: FAS for Part 2 included all participants enrolled in Part 2. Here, N (Overall Number of Participants Analyzed) signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentages of participants
Arm/Group | Part 2: Guselkumab (Week 0-52)
Number analyzed (Participants) | 24
Percentages of participants
  Week 8 | 50.0
  Week 16 | 58.3
  Week 28 | 66.7
  Week 36 | 62.5
  Week 52 | 66.7

22. Secondary Outcome: Part 1: Percentage of Participants With Family Dermatology Life Quality Index (FDLQI) of 0 or 1 at Week 16 Among Participants With a Baseline FDLQI >1
Description: The FDLQI was a 10-item questionnaire that examined the impact of participant's skin disease on different aspects of their QoL (example: emotional, physical well-being, relationships, social life, leisure activities, burden of care, job/study, housework and expenditure) over the last 1 month, as assessed by a family member/partner. Each item had a four-point response option, where Not at all/Not relevant = 0; A little = 1; Quite a lot = 2; and Very much = 3. The scores of individual items (0-3) were added to give a total scale score that ranged from 0 to 30; a higher score indicated greater impairment of QoL.
Time Frame: At Week 16
Population: as for outcome 20
Measure: Number; unit: Percentages of participants
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16)
Number analyzed (Participants) | 23 | 36 | 26
Percentages of participants | 13.0 | 36.1 | 24.0
Statistical Analysis 1: Comparison: Group 1 (Part 1): Placebo (Week 0-16) vs Group 2 (Part 1): Guselkumab (Week 0-16); Guselkumab Vs Placebo; Test type: Superiority; p = 0.139, Fisher Exact — p-value is nominal; [statistical method as in outcome 1, analysis 1]; Difference in Percentage = 23.1, 95% CI 2-sided [-3.4 to 47.0]

23. Secondary Outcome: Part 2: Percentage of Participants With Family Dermatology Life Quality Index (FDLQI) of 0 or 1 Through Week 52 Among Participants With a Baseline FDLQI >1
Description: The FDLQI was a 10-item questionnaire that examine the impact of participant's skin disease on different aspects of their QoL (example, emotional, physical well-being, relationships, social life, leisure activities, burden of care, job/study, housework and expenditure) over the last 1 month, as assessed by a family member/partner. Each item had a four-point response option, where Not at all/Not relevant = 0; A little = 1; Quite a lot = 2; and Very much = 3. The scores of individual items (0-3) were added to give a total scale score that ranged from 0 to 30; a higher score indicates greater impairment of QoL.
Time Frame: Weeks 8, 16, 28, 36, and 52
Population: as for outcome 21
Measure: Number; unit: Percentages of participants
Arm/Group | Part 2: Guselkumab (Week 0-52)
Number analyzed (Participants) | 22
Percentages of participants
  Week 8 | 27.3
  Week 16 | 31.8
  Week 28 | 59.1
  Week 36 | 36.4
  Week 52 | 50.0

24. Secondary Outcome: Part 1: Change From Baseline in FDLQI Score at Week 16
Description: The FDLQI was a 10-item questionnaire that examined the impact of participant's skin disease on different aspects of their QoL (example, emotional, physical well-being, relationships, social life, leisure activities, burden of care, job/study, housework and expenditure) over the last 1 month, as assessed by a family member/partner. Each item had a four-point response option, where Not at all/Not relevant = 0; A little = 1; Quite a lot = 2; and Very much = 3. The scores of individual items (0-3) are added to give a total scale score that ranged from 0 to 30; a higher score indicates greater impairment of QoL.
Time Frame: Baseline and Week 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16)
Number analyzed (Participants) | 24 | 41 | 23
Score on a scale | -0.50 (6.984) | -6.22 (6.299) | -6.22 (4.814)
Statistical Analysis 1: Comparison: Group 1 (Part 1): Placebo (Week 0-16) vs Group 2 (Part 1): Guselkumab (Week 0-16); Guselkumab Vs Placebo; Test type: Superiority; p < 0.001, MMRM model — p-value is nominal; Difference in LS Mean = -5.44, 95% CI 2-sided [-8.00 to -2.87]

25. Secondary Outcome: Part 2: Change From Baseline in FDLQI Score Through Week 52
Description: The FDLQI was a 10-item questionnaire that examine the impact of participant's skin disease on different aspects of their QoL (example, emotional, physical well-being, relationships, social life, leisure activities, burden of care, job/study, housework and expenditure) over the last 1 month, as assessed by a family member/partner. Each item had a four-point response option, where Not at all/Not relevant = 0; A little = 1; Quite a lot = 2; and Very much = 3. The scores of individual items (0-3) are added to give a total scale score that ranged from 0 to 30; a higher score indicated greater impairment of QoL.
Time Frame: Baseline, Weeks 8, 16, 28, 36, and 52
Population: FAS for Part 2 included all participants enrolled in Part 2. Here, N (Overall Number of Participants Analyzed) signifies participants evaluable for this outcome measure and n (number analyzed) signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Part 2: Guselkumab (Week 0-52)
Number analyzed (Participants) | 27
Score on scale
  Week 8 | -5.4 (5.58)
  Week 16: number analyzed (Participants) | 25
  Week 16 | -5.5 (5.90)
  Week 28 | -7.5 (6.15)
  Week 36: number analyzed (Participants) | 26
  Week 36 | -6.7 (5.00)
  Week 52: number analyzed (Participants) | 26
  Week 52 | -7.8 (5.68)

26. Secondary Outcome: Part 1: Change From Baseline in Body Surface Area (BSA) With Psoriasis Skin Involvement at Week 16
Description: Change from baseline in percent body surface area with psoriasis skin involvement was reported. BSA as physical measure to define disease severity is to determine how much of the BSA is affected by psoriasis. Involved BSA is calculated by using the palm of the participant's hand as equivalent to 1% of the BSA (rule of palm). Psoriasis affected BSA under 5% suggests mild psoriasis, a BSA of 5% to 10% is considered moderate, and an involved BSA of over 10% indicates severe psoriasis.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group 1 (Part 1): Placebo (Week 0-16) | Group 2 (Part 1): Guselkumab (Week 0-16) | Group 3 (Part 1): Etanercept (Week 0-16)
Number analyzed (Participants) | 25 | 41 | 24
Units on a scale | -2.84 (13.861) | -19.59 (17.645) | -17.50 (10.628)
Statistical Analysis 1: Comparison: Group 1 (Part 1): Placebo (Week 0-16) vs Group 2 (Part 1): Guselkumab (Week 0-16); Guselkumab Vs Placebo; Test type: Superiority; p < 0.001, MMRM model — p-value is nominal; LS Mean difference = -14.78, 95% CI 2-sided [-20.28 to -9.28]

27. Secondary Outcome: Parts 2: Change From Baseline in BSA With Psoriasis Skin Involvement Over Time Through Week 52
Description: as for outcome 26
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 28, 36, 44, and 52
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part 2: Guselkumab (Week 0-52)
Number analyzed (Participants) | 28
Units on a scale
  Week 4 | -6.9 (7.94)
  Week 8 | -16.8 (12.00)
  Week 12: number analyzed (Participants) | 27
  Week 12 | -19.6 (12.58)
  Week 16: number analyzed (Participants) | 26
  Week 16 | -22.7 (13.57)
  Week 20: number analyzed (Participants) | 27
  Week 20 | -24.0 (13.46)
  Week 28: number analyzed (Participants) | 27
  Week 28 | -26.0 (14.61)
  Week 36 | -26.3 (14.42)
  Week 44: number analyzed (Participants) | 27
  Week 44 | -26.5 (14.05)
  Week 52: number analyzed (Participants) | 27
  Week 52 | -26.4 (14.52)

28. Secondary Outcome: LTE Phase: Percentage of Participants Who Achieved PASI Responses (PASI 50, 75, 90, and 100) Over Time
Time Frame: From Week 52 to End of the study (EOS) (December 2026)
Reporting Status: Not Posted, anticipated posting 2027-12

29. Secondary Outcome: LTE Phase: Percentage of Participants Who Achieved IGA Score of (Cleared [0], Cleared [0] or Minimal [1], Mild or Better [<=2] Over Time
Time Frame: From Week 52 to EOS (December 2026)
Reporting Status: Not Posted, anticipated posting 2027-12

30. Secondary Outcome: LTE Phase: Percent Improvement From Baseline in PASI Over Time
Time Frame: From Week 52 to EOS (December 2026)
Reporting Status: Not Posted, anticipated posting 2027-12

31. Secondary Outcome: LTE Phase: Change From Baseline in BSA With Psoriasis Skin Involvement Over Time
Time Frame: From Week 52 to EOS (Dec 2026)
Reporting Status: Not Posted, anticipated posting 2027-12

32. Secondary Outcome: LTE Phase: Percentage of Participants Who Achieved PASI Responses (PASI 50, 75, 90,and 100) at Weeks 60 and 84 After Retreatment Among Guselkumab Participants Who Were Withdrawn From Guselkumab at Week 16 and Retreated Upon Loss of Response or at Week 52
Time Frame: Week 60 and Week 84
Reporting Status: Not Posted, anticipated posting 2027-12

33. Secondary Outcome: LTE Phase: Percentage of Participants Who Achieved IGA Score of (Cleared [0], Cleared [0] or Minimal [1], Mild or Better [<=2] at Weeks 60 and 84 After Retreatment
Time Frame: Week 60 and Week 84
Reporting Status: Not Posted, anticipated posting 2027-12

34. Secondary Outcome: LTE Phase: Percent Improvement in PASI Responses (PASI 50, 75, 90, and 100) at Weeks 60 and 84 After Retreatment Among Guselkumab Subjects Who Were Withdrawn From Guselkumab at Week 16 and Subsequently Retreated Upon Loss of Response or at Week 52
Time Frame: Week 60 and Week 84
Reporting Status: Not Posted, anticipated posting 2027-12

35. Secondary Outcome: LTE Phase: Change From Baseline in BSA at Weeks 60 and 84 After Retreatment Among Guselkumab Subjects Who Were Withdrawn From Guselkumab at Week 16 and Subsequently Retreated Upon Loss of Response or at Week 52
Time Frame: Week 60 and Week 84
Reporting Status: Not Posted, anticipated posting 2027-12

ADVERSE EVENTS:
Time Frame: PCP (Part 1): Week 0 to 16; Withdrawal and re-treatment period (Part 1): Week 16 to 52; Part 2: Week 0 to 52
Description: Safety analysis set included all treated participants who received at least 1 injection of study agent (partial or complete). As planned, data for Part 2 has been reported collectively from Week 0 to 52 since participants continued the same treatment through Week 52.
Groups:
- PCP-Group 1 (Part 1): Placebo (Week 0-16): Adolescent participants (aged >=12 to <18 years) received placebo matched to guselkumab as subcutaneous (SC) injection at Weeks 0, 4, and 12 during the placebo-controlled period (PCP). Once adolescent participants completed Week 16, eligible participants aged >=6 to <12 years were enrolled and began receiving the same dose regimen starting from Week 0 until Week 16.
- PCP-Group 2 (Part 1): Guselkumab (Week 0-16): Adolescent participants received weight-adjusted doses of guselkumab (1.3 mg/kg for body weight [BW] <70 kg, 100 mg for BW >=70 kg) via subcutaneous injection at Weeks 0, 4, and 12 during PCP. Once adolescent participants completed Week 16, eligible participants aged >=6 to <12 years began receiving the same dose regimen starting from Week 0 until Week 16.
- PCP-Group 3 (Part 1): Etanercept (Week 0-16): Adolescent participants received weight-based dose of open-label etanercept 0.8 mg/kg for BW <63 kg and 50 mg for BW >=63 kg SC injection once weekly from Week 0 to Week 15. Once adolescent participants completed Week 16, eligible participants aged >=6 to <12 years began receiving the same dose regimen starting from Week 0 until Week 16.
- Withdrawal and Re-treatment Period-Group 1 (Part 1): Placebo to Guselkumab (Week 16-52): Participants who received placebo during PCP were assessed for psoriasis area and severity index (PASI) response at Week 16. Participants who were PASI 90 non-responders at Week 16 received weight-based doses of guselkumab (1.3 mg/kg for BW <70 kg, 100 mg for BW >=70 kg) as SC injection at Weeks 16, 20 and then every 8 weeks (q8w) thereafter through Week 52. Participants who were PASI 90 responders at Week 16 stopped treatment until they lost >= 50 percent (%) of their Week 16 PASI response, at which time they were treated with guselkumab 1.3 mg/kg or 100 mg depending on their body weight followed by a dose 4 weeks later, and then guselkumab q8w thereafter through Week 52. All participants who completed Part 1 of the main study through Week 52 were offered the opportunity to participate in an open-label LTE.
- Withdrawal and Re-treatment Period-Group 2 (Part 1): Guselkumab (Week 16-52): Participants who received guselkumab during PCP were assessed for PASI response at Week 16. Participants who were PASI 90 non-responders at Week 16 received weight-based doses of guselkumab (1.3 mg/kg for BW <70 kg, 100 mg for BW >=70 kg) as SC injection at Weeks 16, 20 and then q8w thereafter through Week 52. Participants who were PASI 90 responders at Week 16 stopped treatment until they lost >= 50 % of their Week 16 PASI response, at which time they were retreated with guselkumab 1.3 mg/kg or 100 mg depending on their body weight followed by a dose 4 weeks later, and then guselkumab every 8 weeks thereafter through Week 52. All participants who completed Part 1 of the main study through Week 52 were offered the opportunity to participate in an open-label LTE.
- Withdrawal and Re-treatment Period- Group 3 (Part 1): Etanercept to Guselkumab (Week 16-52): Participants who received etanercept during the PCP had the option to continue in the study or to discontinue the study. Participants that continued received weight-based doses of guselkumab (1.3 mg/kg for body weight [BW] <70 kg, 100 mg for BW >=70 kg) as SC injection at Weeks 20 and 24, followed by q8w dosing through Week 48 and remaining participants discontinued from the study. All participants who completed Part 1 of the main study through Week 52 were offered the opportunity to participate in an open-label LTE.
Arm/Group | PCP-Group 1 (Part 1): Placebo (Week 0-16) | PCP-Group 2 (Part 1): Guselkumab (Week 0-16) | PCP-Group 3 (Part 1): Etanercept (Week 0-16) | Withdrawal and Re-treatment Period-Group 1 (Part 1): Placebo to Guselkumab (Week 16-52) | Withdrawal and Re-treatment Period-Group 2 (Part 1): Guselkumab (Week 16-52) | Withdrawal and Re-treatment Period- Group 3 (Part 1): Etanercept to Guselkumab (Week 16-52) | Part 2: Guselkumab (Week 0-52)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/41 | 0/26 | 0/23 | 0/41 | 0/22 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/41 | 0/26 | 1/23 | 0/41 | 0/22 | 1/28
Other Adverse Events (participants affected / at risk) | 17/25 | 17/41 | 15/26 | 16/23 | 29/41 | 13/22 | 23/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PCP-Group 1 (Part 1): Placebo (Week 0-16) (N=25) | PCP-Group 2 (Part 1): Guselkumab (Week 0-16) (N=41) | PCP-Group 3 (Part 1): Etanercept (Week 0-16) (N=26) | Withdrawal and Re-treatment Period-Group 1 (Part 1): Placebo to Guselkumab (Week 16-52) (N=23) | Withdrawal and Re-treatment Period-Group 2 (Part 1): Guselkumab (Week 16-52) (N=41) | Withdrawal and Re-treatment Period- Group 3 (Part 1): Etanercept to Guselkumab (Week 16-52) (N=22) | Part 2: Guselkumab (Week 0-52) (N=28)
Chronic Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PCP-Group 1 (Part 1): Placebo (Week 0-16) (N=25) | PCP-Group 2 (Part 1): Guselkumab (Week 0-16) (N=41) | PCP-Group 3 (Part 1): Etanercept (Week 0-16) (N=26) | Withdrawal and Re-treatment Period-Group 1 (Part 1): Placebo to Guselkumab (Week 16-52) (N=23) | Withdrawal and Re-treatment Period-Group 2 (Part 1): Guselkumab (Week 16-52) (N=41) | Withdrawal and Re-treatment Period- Group 3 (Part 1): Etanercept to Guselkumab (Week 16-52) (N=22) | Part 2: Guselkumab (Week 0-52) (N=28)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Conjunctivitis Allergic (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Myopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Application Site Haematoma (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1
Influenza Like Illness (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Injection Site Erythema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Injection Site Haematoma (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Injection Site Induration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection Site Pruritus (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection Site Swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 1
Seasonal Allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Bacterial Vulvovaginitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 1 | 0
Chronic Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 6
Ear Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterobiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gastrointestinal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Helminthic Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lice Infestation (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Molluscum Contagiosum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 7 | 5 | 3 | 8 | 9 | 4 | 7
Otitis Externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis Media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 1 | 2 | 1 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Tinea Capitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinea Versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 4 | 2 | 0 | 6 | 3 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral Diarrhoea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peroneal Nerve Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Glucose Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Pressure Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac Murmur (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver Function Test Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
White Blood Cell Count Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ligament Laxity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 3 | 1 | 2 | 3 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Attention Deficit Hyperactivity Disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 3
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diffuse Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lichen Planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT03451851/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT03451851/SAP_001.pdf